CLINICAL TRIAL: NCT06300619
Title: Evaluating the Impact of Introducing the 4-quadrant Stability Model Into Pilates Instruction: Effects on Function Among Adults With Multiple Sclerosis
Brief Title: Pilates+4MS: Pilates Intervention for Multiple Sclerosis
Acronym: P+4MS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Colorado Springs (Other)
Collaborators: University of Illinois at Urbana-Champaign (Other)
Responsible Party: Principal Investigator, Brynn Adamson, Assistant Professor, University of Colorado, Colorado Springs
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2022-066
Record Dates: First submitted 2024-01-12; First posted 2024-03-08 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Exercise Movement Techniques

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants know that there are 2 Pilates groups, but not which group is under investigation vs. the comparison group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pilates (Active Comparator): Standard Pilates Protocol with no hip/shoulder cuff cuing. Delivered from a seated position.
  Interventions: Behavioral: Pilates
- Pilates+4 (Experimental): Pilates protocol that involves hip and shoulder cuff activation and stabilization exercises and cues to augment the Pilates exercise.
  Interventions: Behavioral: Pilates+4

INTERVENTIONS:
Behavioral: Pilates+4 — 12 weeks of seated Pilates twice weekly. In weeks 1-3, participants receive training on hip and shoulder cuff activation. This occurs through active isometric pressure on the stabilizing limb (not the moving limb during a Pilates movement) for 3 seconds at 30% strength using the participants' own hand (e.g., pressure on the outside of the knee with knee pressing against hand) prior to engaging in each exercise. Following the first 3 weeks, participants in the Pilates+4 group engage in the same Pilates protocol as the comparator group, however, they receive 4-quadrant cues for hip and shoulder cuff activation as they learned in weeks 1-3.
  Arms: Pilates+4
Behavioral: Pilates — 12 weeks of seated Pilates twice weekly. 18 exercises standard in Pilates instruction will be provided with standard Pilates cues (i.e., core activation, cuing the moving limb, breathing synchronization).
  Arms: Pilates

SUMMARY:
The goal of this clinical trial is to test the physical health benefits of seated Pilates in the multiple sclerosis (MS) population. The main questions it aims to answer are: 1) is it feasible to deliver a seated Pilates class for 12 weeks, twice weekly over Zoom in a group format among participants with mild, moderate, and severe multiple sclerosis? 2) what are the mobility, balance, and symptom benefits of a 12-week seated Pilates class? 3) Does incorporating hip and shoulder stabilization augment the benefits compared to a standard seated Pilates protocol? 4) Are there benefits to physical activity participation? Participants will be screened over the phone for eligibility criteria and then scheduled for in-person data collection. In person data collection will involve: 1) completing the Timed 25-Foot Walk a total of 4 times, 2) the Timed Up and Go a total of 4 times, 3) the Berg Balance Scale a total of 2 times, and 4) a set of 8 questionnaires about multiple sclerosis symptoms and impact, and physical activity behavior. Participants will receive a FitBit and then will be randomized into the Pilates only group or the Pilates+4-Quadrant stability group for the intervention. The intervention is 12 weeks long, both groups meet twice weekly on Zoom for 60 minutes with 1 of 2 instructors and other class participants (12 per group). They wear the FitBit for all 12 weeks and then return for testing to repeat testing items 1-4 above. Researchers will compare the functional outcomes between the Pilates only group and the Pilates+4-Quadrant Stability group to see if there are differences in mobility, balance and physical activity outcomes.

DETAILED DESCRIPTION:
Twenty-four persons with mild, moderate, and severe MS (PwMS) will be recruited and screened for eligibility criteria. The investigators will actively recruit PwMS through local MS support group events, and previous participant databases. Interested participants will be screened for inclusion/exclusion criteria, i.e. aged 18+, diagnosis of MS, relapse-free in the past 30 days, access to a computer/tablet with internet, willingness to participate in an exercise program, Physical Activity Readiness Questionnaire <2 affirmatives, between 3 and 5 on Patient Determined Disease Steps (PDDS 3-5). Participants who are qualified will be invited to take part in the study.

The participant involvement includes 4 main components. First, participants will be asked to complete a 90-minute testing session at the Hybl Building on the University of Colorado Colorado Springs (UCCS) campus. This testing session will involve some balance and walking tests (Berg Balance Scale, Timed Up and Go and Timed 25-foot walk) and completion of several questionnaires (Multiple Sclerosis Impact Scale, Late Life Function and Disability Index, Godin Leisure Time Exercise Questionnaire, Leeds Multiple Sclerosis Quality of Life Scale, Modified Fatigue Impact Scales, and Self-Reported Expanded Disability Status Scale). After filling out the questionnaires, participants will repeat the balance and walking tests but with cues mirroring the cues that will be given in the 4-quadrant group (stabilize prior to beginning the movement). Participants will wear an E4 activity monitor (small device worn like a watch) while completing these tasks and investigators will video record the balance and walking tests for later movement analysis.

Upon completion of pre-intervention (T1) tests participants will be randomized into either the Pilates only or the Pilates+ (4-quadrant stability) groups. The participants will be given a manual based on their group assignment with information about using Zoom, class schedule, safety tips, and how-to guides to complete the exercises. The 4-quadrant group will have additional information about functional movement which the other group will only receive upon completion of the intervention. The investigators will also provide participants with a resistance band (TheraBand) and two yoga blocks for them to use while in the study. Participants will be allowed to keep the equipment afterwards. The investigators will instruct participants on the use of a physical activity monitor (FitBit) and help them download an app to allow them to track their physical activity data and send it to the team. The FitBit will be returned upon completion of the study.

The second part of the study involves having the participant wearing the FitBit monitor and sharing their physical activity participation with the team for a period of 12 weeks.

The third part of the study involves participating in a 12-week Pilates program that will be held twice a week for 60 minutes on Zoom. The classes will be seated and taught by trained Pilates instructors with extensive training and knowledge of MS. Aside from the instructor being present, a member of the research team will also always be present to provide technical troubleshooting support, answer questions and watch the participants and alert the instructor of unsafe practices. Participants in the Pilates only class will participate in 24 sessions of Pilates with standard Pilates cues and movements. Participants in the Pilates+ 4 quadrant group will begin with 6 sessions of functional exercise helping them to learn the 4-quadrant stability cues in their bodies (hip and shoulder activation, eye-tracking etc.) Then, this group will transition to the same Pilates protocol as the first group but will continue to receive 4-quadrant cues. In both classes, all exercises will be demonstrated from a seated position.

The fourth part of the study involves returning to UCCS campus for another 90-minute testing session where participants will repeat the balance and walking tests as well as the questionnaires. At the last testing session participants will receive one additional survey - a feedback survey on the program.

All data will be analyzed using Statistical Package for Social Science (SPSS) Statistics 29.0 (Chicago, IL).

ELIGIBILITY:
Inclusion Criteria:

* aged 18+
* diagnosis of MS (self-reported)
* relapse-free in the past 30 days
* access to a computer/tablet with internet
* willingness to participate in a 12-week exercise program
* Physical Activity Readiness Questionnaire (PARQ) <2 affirmatives.

Exclusion Criteria:

* aged <18
* relapse in past 30 days
* PARQ 2+ affirmatives

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2022-04-05 (Actual); Primary Completion 2022-08-25 (Actual); Study Completion 2022-08-25 (Actual)

PRIMARY OUTCOMES:
Timed 25 Foot Walk | Immediately pre intervention (within 2 weeks before the intervention) and immediately post intervention (within 2 weeks following the last date of the intervention)
  Participants are instructed to walk 25 feet as fast as they can in the limits of their safety. This is timed.
Timed Up and Go | Immediately pre intervention (within 2 weeks before the intervention) and immediately post intervention (within 2 weeks following the last date of the intervention)
  Participants begin the test in a seated position. There is a mark on the floor 10 feet from the edge of their seat. When the tester says go, the participant stands from their seat, walks at their normal, comfortable, every-day walking pace to the mark, turns around, walks back to the chair, and sits down again. This is timed.
Berg Balance Scale | Immediately pre intervention (within 2 weeks before the intervention) and immediately post intervention (within 2 weeks following the last date of the intervention)
  This is a 14-item balance battery involving static and dynamic balance challenges. Each challenge is scored by the tester based on the participants' performance and the total is calculated. The scores range from 0 to 56 with a higher score indicating better functional balance.

SECONDARY OUTCOMES:
Triaxial Accelerometer (FitBit) Physical Activity Data (minutes of wear time in sedentary time and light, moderate and vigorous physical activity) | 12 weeks of daily wearing.
  Each participant receives a FitBit Inspire device (wearable physical activity monitor worn on the wrist) which measures daily physical activity behavior.
The Godin-Shepherd Leisure Time Exercise Questionnaire | Immediately pre intervention (within 2 weeks before the intervention) and immediately post intervention (within 2 weeks following the last date of the intervention)
  This is a survey of 4 items asking about light, moderate, and high intensity exercise behavior as well as one question on how many times per week the participant is active enough to sweat. The values range from 0 to 119 with higher scores equating to increased physical activity participation.
Late-Life Function and Disability Instrument Short Form | Immediately pre intervention (within 2 weeks before the intervention) and immediately post intervention (within 2 weeks following the last date of the intervention)
  This survey is a measure of function and disability/impairment. The scale scoring ranges from 0-100 with higher scores indicating increased function and lower impact of disability on daily activity.
Leeds Multiple Sclerosis Quality of Life Scale | Immediately pre intervention (within 2 weeks before the intervention) and immediately post intervention (within 2 weeks following the last date of the intervention)
  This scale measures subjective quality of life. The scale scores range from 0-24 with higher scores indicating improved quality of life.
Modified Fatigue Impact Scale | Immediately pre intervention (within 2 weeks before the intervention) and immediately post intervention (within 2 weeks following the last date of the intervention)
  This scale measures the perceptions that fatigue impacts various aspects of the participants activities of daily living and participation. The scores range from 0-36 with higher scores indicating worse fatigue impact.
Multiple Sclerosis Impact Scale | Immediately pre intervention (within 2 weeks before the intervention) and immediately post intervention (within 2 weeks following the last date of the intervention)
  This scale measures the subjective perception of how MS impacts various aspects of the participants activities of daily living and participation across physical and psychological components. This scale has two subscales (physical and psychological). Scores on the physical impact scale can range from 20 to 80 and on the psychological impact scale from 9 to 36, with lower scores indicating little impact of MS and higher scores indicating greater impact.

CONTACTS AND LOCATIONS:
Locations (1):
- Hybl Sports Medicine and Performance Center, Colorado Springs, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ensari I, Motl RW, McAuley E. Structural and construct validity of the Leeds Multiple Sclerosis Quality of Life scale. Qual Life Res. 2016 Jun;25(6):1605-11. doi: 10.1007/s11136-015-1202-5. Epub 2015 Dec 11. PMID 26660145
- [Background] Arain M, Campbell MJ, Cooper CL, Lancaster GA. What is a pilot or feasibility study? A review of current practice and editorial policy. BMC Med Res Methodol. 2010 Jul 16;10:67. doi: 10.1186/1471-2288-10-67. PMID 20637084
- [Background] Downs S. The Berg Balance Scale. J Physiother. 2015 Jan;61(1):46. doi: 10.1016/j.jphys.2014.10.002. Epub 2014 Dec 1. No abstract available. PMID 25476663
- [Background] Cattaneo D, Jonsdottir J, Repetti S. Reliability of four scales on balance disorders in persons with multiple sclerosis. Disabil Rehabil. 2007 Dec 30;29(24):1920-5. doi: 10.1080/09638280701191859. Epub 2007 Apr 26. PMID 17852286
- [Background] Decavel P, Moulin T, Sagawa Y Jr. Gait tests in multiple sclerosis: Reliability and cut-off values. Gait Posture. 2019 Jan;67:37-42. doi: 10.1016/j.gaitpost.2018.09.020. Epub 2018 Sep 22. PMID 30269001
- [Background] Donoghue D; Physiotherapy Research and Older People (PROP) group; Stokes EK. How much change is true change? The minimum detectable change of the Berg Balance Scale in elderly people. J Rehabil Med. 2009 Apr;41(5):343-6. doi: 10.2340/16501977-0337. PMID 19363567
- [Background] Duff WRD, Andrushko JW, Renshaw DW, Chilibeck PD, Farthing JP, Danielson J, Evans CD. Impact of Pilates Exercise in Multiple Sclerosis: A Randomized Controlled Trial. Int J MS Care. 2018 Mar-Apr;20(2):92-100. doi: 10.7224/1537-2073.2017-066. PMID 29670495
- [Background] Haley SM, Jette AM, Coster WJ, Kooyoomjian JT, Levenson S, Heeren T, Ashba J. Late Life Function and Disability Instrument: II. Development and evaluation of the function component. J Gerontol A Biol Sci Med Sci. 2002 Apr;57(4):M217-22. doi: 10.1093/gerona/57.4.m217. PMID 11909886
- [Background] Heesen C, Bohm J, Reich C, Kasper J, Goebel M, Gold SM. Patient perception of bodily functions in multiple sclerosis: gait and visual function are the most valuable. Mult Scler. 2008 Aug;14(7):988-91. doi: 10.1177/1352458508088916. Epub 2008 May 27. PMID 18505775
- [Background] Kaufmann M, Salmen A, Barin L, Puhan MA, Calabrese P, Kamm CP, Gobbi C, Kuhle J, Manjaly ZM, Ajdacic-Gross V, Schafroth S, Bottignole B, Ammann S, Zecca C, D'Souza M, von Wyl V; Swiss Multiple Sclerosis Registry (SMSR). Development and validation of the self-reported disability status scale (SRDSS) to estimate EDSS-categories. Mult Scler Relat Disord. 2020 Jul;42:102148. doi: 10.1016/j.msard.2020.102148. Epub 2020 Apr 28. PMID 32371376
- [Background] Kinnett-Hopkins D, Adamson B, Rougeau K, Motl RW. People with MS are less physically active than healthy controls but as active as those with other chronic diseases: An updated meta-analysis. Mult Scler Relat Disord. 2017 Apr;13:38-43. doi: 10.1016/j.msard.2017.01.016. Epub 2017 Feb 1. PMID 28427699
- [Background] Lancaster GA. Pilot and feasibility studies come of age! Pilot Feasibility Stud. 2015;1(1):1. doi: 10.1186/2055-5784-1-1. Epub 2015 Jan 12. PMID 29611687
- [Background] Learmonth YC, Dlugonski DD, Pilutti LA, Sandroff BM, Motl RW. The reliability, precision and clinically meaningful change of walking assessments in multiple sclerosis. Mult Scler. 2013 Nov;19(13):1784-91. doi: 10.1177/1352458513483890. Epub 2013 Apr 15. PMID 23587605
- [Background] Learmonth YC, Paul L, McFadyen AK, Mattison P, Miller L. Reliability and clinical significance of mobility and balance assessments in multiple sclerosis. Int J Rehabil Res. 2012 Mar;35(1):69-74. doi: 10.1097/MRR.0b013e328350b65f. PMID 22315143
- [Background] Marques KAP, Trindade CBB, Almeida MCV, Bento-Torres NVO. Pilates for rehabilitation in patients with multiple sclerosis: A systematic review of effects on cognition, health-related physical fitness, general symptoms and quality of life. J Bodyw Mov Ther. 2020 Apr;24(2):26-36. doi: 10.1016/j.jbmt.2020.01.008. Epub 2020 Feb 6. PMID 32507148
- [Background] Motl RW, Bollaert RE, Sandroff BM. Validation of the Godin Leisure-Time Exercise Questionnaire classification coding system using accelerometry in multiple sclerosis. Rehabil Psychol. 2018 Feb;63(1):77-82. doi: 10.1037/rep0000162. Epub 2017 Jul 31. PMID 28758772
- [Background] Motl RW, Cohen JA, Benedict R, Phillips G, LaRocca N, Hudson LD, Rudick R; Multiple Sclerosis Outcome Assessments Consortium. Validity of the timed 25-foot walk as an ambulatory performance outcome measure for multiple sclerosis. Mult Scler. 2017 Apr;23(5):704-710. doi: 10.1177/1352458517690823. Epub 2017 Feb 16. PMID 28206828
- [Background] Oliver GD, Washington JK, Barfield JW, Gascon SS, Gilmer G. Quantitative Analysis of Proximal and Distal Kinetic Chain Musculature During Dynamic Exercises. J Strength Cond Res. 2018 Jun;32(6):1545-1553. doi: 10.1519/JSC.0000000000002036. PMID 29786622
- [Background] Paltamaa J, Sarasoja T, Leskinen E, Wikstrom J, Malkia E. Measures of physical functioning predict self-reported performance in self-care, mobility, and domestic life in ambulatory persons with multiple sclerosis. Arch Phys Med Rehabil. 2007 Dec;88(12):1649-57. doi: 10.1016/j.apmr.2007.07.032. PMID 18047881
- [Background] Riazi A, Hobart JC, Lamping DL, Fitzpatrick R, Thompson AJ. Multiple Sclerosis Impact Scale (MSIS-29): reliability and validity in hospital based samples. J Neurol Neurosurg Psychiatry. 2002 Dec;73(6):701-4. doi: 10.1136/jnnp.73.6.701. PMID 12438473
- [Background] Rodriguez-Fuentes G, Silveira-Pereira L, Ferradans-Rodriguez P, Campo-Prieto P. Therapeutic Effects of the Pilates Method in Patients with Multiple Sclerosis: A Systematic Review. J Clin Med. 2022 Jan 28;11(3):683. doi: 10.3390/jcm11030683. PMID 35160134
- [Background] Sanchez-Lastra MA, Martinez-Aldao D, Molina AJ, Ayan C. Pilates for people with multiple sclerosis: A systematic review and meta-analysis. Mult Scler Relat Disord. 2019 Feb;28:199-212. doi: 10.1016/j.msard.2019.01.006. Epub 2019 Jan 3. PMID 30623859
- [Background] Sebastiao E, Sandroff BM, Learmonth YC, Motl RW. Validity of the Timed Up and Go Test as a Measure of Functional Mobility in Persons With Multiple Sclerosis. Arch Phys Med Rehabil. 2016 Jul;97(7):1072-7. doi: 10.1016/j.apmr.2015.12.031. Epub 2016 Mar 2. PMID 26944709
- [Background] van der Linden ML, Bulley C, Geneen LJ, Hooper JE, Cowan P, Mercer TH. Pilates for people with multiple sclerosis who use a wheelchair: feasibility, efficacy and participant experiences. Disabil Rehabil. 2014;36(11):932-9. doi: 10.3109/09638288.2013.824035. Epub 2013 Aug 19. PMID 23957639